CLINICAL TRIAL: NCT06925321
Title: An Interventional Phase 3, Open-label, Two-cohort Study to Investigate the Efficacy and Safety of Fosmanogepix in Adult Patients With Invasive Mold Infections Caused by Aspergillus Spp., Fusarium Spp., Lomentospora Prolificans, Mucorales Fungi, or Other Multidrug Resistant Molds
Brief Title: A Phase 3 Efficacy and Safety Study of Fosmanogepix for the Treatment of Adult Patients With Invasive Mold Infections.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMGX-CS-302
Expanded Access: NCT06433128 (Available)
Record Dates: First submitted 2025-03-27; First posted 2025-04-13 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Invasive Mold Infections
Keywords: Fungal infection; Antifungal; Mold infection; Rare molds; Multidrug resistant mold; Aspergillus spp.; Fusarium spp.; Lomentospora prolificans; Mucorales fungi; Scedosporium spp.
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Intervention Model Description: An open-label, 2-cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: Experimental Treatment (Experimental): Patients will receive the study drug.
  Fosmanogepix will be administered as an Intravenous (IV) infusion or in oral form.
  Interventions: Drug: Fosmanogepix IV infusion; Drug: Fosmanogepix oral tablet
- Cohort A: Comparator Antifungal Treatment (Active Comparator): Best available therapy (BAT) administered as IV or orally per standard guidelines.
  Interventions: Drug: Standard of care antifungal therapy
- Cohort B (Experimental): Patients will receive the study drug.
  Fosmanogepix will be administered as an Intravenous (IV) infusion or in oral form.
  Interventions: Drug: Fosmanogepix IV infusion; Drug: Fosmanogepix oral tablet

INTERVENTIONS:
Drug: Fosmanogepix IV infusion — Fosmanogepix will be administered IV
  Arms: Cohort A: Experimental Treatment; Cohort B
Drug: Standard of care antifungal therapy — Standard of care antifungal therapy will be administered in accordance with their respective product labels and/or standard practice guidelines
  Arms: Cohort A: Comparator Antifungal Treatment
Drug: Fosmanogepix oral tablet — Fosmanogepix will be administered orally.
  Arms: Cohort A: Experimental Treatment; Cohort B

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of fosmanogepix (administered IV or oral) for the treatment of adult patients with invasive mold infections. The study is looking for patients who have been diagnosed with invasive mold infections. The maximum study duration will be approximately 8 months, including a target study treatment duration of 84 days which can be extended up to 180 days and follow-up period.

The patient will be assigned to one of two treatment cohorts:

Cohort A (primary therapy): Patients will receive either the study drug or institutional standard of care antifungal treatment.

Cohort B (salvage treatment; i.e. treatment given after patients did not respond to previous treatments or did not tolerate them): Patients will receive the study drug

The primary aim is to compare the all cause mortality with a fixed threshold at Day 42.

ELIGIBILITY:
Main Inclusion Criteria:

1. Diagnosis of proven or probable Invasive mold infection (IMI) defined in accordance with the Revision and Update of the Consensus Definitions of Invasive Fungal Disease from the EORTC/MSGERC as adapted for this study and caused by Aspergillus spp. (in patients with limited treatment options), Fusarium spp., Lomentospora prolificans, Mucorales fungi, or other multi-drug resistant molds.
2. Patient's condition allows for appropriate infection source control measures.

Main Exclusion Critera:

1. Refractory hematologic malignancy.
2. Chronic aspergillosis, aspergilloma, or allergic bronchopulmonary aspergillosis.
3. COVID-19 associated mucormycosis.
4. Invasive fungal disease caused by more than one fungal pathogen is not permitted in Cohort A but is permitted in Cohort B.
5. Patients with a Karnofsky Performance Status < 20 at Screening.
6. Requirement, or anticipated requirement, for hemodialysis, peritoneal dialysis, or hemofiltration.
7. Patients with known human immunodeficiency virus infection.
8. Ongoing neurological disorders.
9. Patients receiving hospice/comfort care only.
10. Other medical or psychiatric condition.
11. Current use of any prohibited concomitant medication(s).
12. Current/ previous administration of an investigational drug within 30 days.
13. Prior enrollment in this or any previous study of fosmanogepix.
14. Moderate or severe hepatic impairment.
15. Patient who is pregnant or lactating.
16. Known hypersensitivity to fosmanogepix, manogepix, or any of their excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Day 42 all-cause mortality rate | Day 42

SECONDARY OUTCOMES:
Proportion of patients with overall response of treatment success | Day 42, Day 84 and up to 180 days
Proportion of patients with clinical response of treatment success | Day 42, Day 84 and up to 180 days
Proportion of patients with mycological response of eradication or presumed eradication | Day 42, Day 84 and up to 180 days
Proportion of patients with radiological response of complete response or partial response | Day 42, Day 84 and up to 180 days
All-cause mortality rate at Day 84 | Day 84
Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), treatment-related AEs, adverse events of special interest (AESI), and AEs leading to discontinuation | Screening up to follow-up 6 weeks after EOST (target duration approximately up to 8 months)
Number of patients with clinically significant laboratory abnormalities | Up to follow-up 6 weeks after EOST (target duration approximately up to 8 months)
Number of patients with abnormal neurological examination findings | Up to follow-up 6 weeks after EOST (target duration approximately up to 8 months)
Assessment of 12-lead electrocardiogram corrected QT (Fridericia method) Interval (ECG QTcF Interval) | Up to follow-up 6 weeks after EOST (target duration approximately up to 8 months)
Plasma concentrations versus time of fosmanogepix (prodrug) and manogepix (active moiety) following IV administration | Pre-dose, 3,6, and 9 hours post-start of the 3-hour IV infusion on Day 3, and at 24 hours (prior to Day 4 dosing)
Plasma concentrations versus time of fosmanogepix (prodrug) and manogepix (active moiety) following oral administration | On days 7, 14, 28, and 42. Post-dose plasma samples will also be collected: 72 hrs and 192 hrs after last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Ionescu, MD, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (18):
- United States (8):
  - University of Alabama at Birmingham School of Medicine, Department of Medicine, Birmingham, Alabama
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Karmanos Cancer Institute - Detroit, Detroit, Michigan
  - University of Minnesota, M Health Fairview Medical Center, Minneapolis, Minnesota
  - Washington University School of Medicine, Infectious Diseases Clinical Research Unit, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Duke Infectious Diseases, Durham, North Carolina
  - The University of Texas Health Science Center at Houston, Department of Internal Medicine, Houston, Texas
- Princess Alexandra Hospital, Woolloongabba, Australia
- Kepler University Hospital GmbH, Department of Internal Medicine IV - Pulmonology, Linz, Austria
- Israel (4):
  - Rambam Health Care Campus, Institute of Infectious Diseases, Haifa
  - Chaim Sheba Medical Center, Department of Infectious Diseases, Ramat Gan
  - The Tel Aviv Sourasky Medical Center, Infectious Diseases Unit, Tel Aviv
  - Shamir Medical Center, Department of Infectious Diseases, Ẕerifin
- Thailand (4):
  - Faculty of Medicine, Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Songklanagarind Hospital, Hat Yai
  - Srinagarind Hospital, Khon Kaen